CLINICAL TRIAL: NCT02691780
Title: Study to Evaluate the Safety and Efficacy of Sorafenib, in Subject With Refractory Solid Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not enrolled
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-02-097
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — Sorafenib

ARMS (1):
- Sorafenib (Experimental): Sorafenib 200mg bid will be administered orally daily every 3weeks
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib
  Other Names: Nexavar

SUMMARY:
This study is a single arm, pilot study of Sorafenib in patient with BRAF mutation Refractory solid tumor and specific sensitivity to Sorafenib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.

To investigate the efficacy and safety of Sorafenib in patient with Refractory solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Provision of fully informed consent prior to study specific procedures.
* Patients must be >= 19 years of age
* BRAF mutation, Refractory solid tumor and/or specific sensitivity to Sorafenib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.
* ECOG Performance status0-2
* Have measurable or evaluated disease based on RECIST 1.1 as determined by investigator.
* Adequate Organ Function Laboratory values

  * Absolute neutrophil count >= 1.5 x 109/L, Hemoglobin >= 9g/dL, Platelets>=100x 109/L Bilirubin <= 1.5 x upper limit of normal AST/ALT <= 2.5 X upper limit of normal(5.0 x upper limit of normal, for subject with liver metastases) Creatinine<= 1.5 X UNL
* Patients of child-bearing potential should be using adequate contraceptive measures should not be breast feeding and must have a negative pregnancy test prior to start of dosing
* Adequate heart function

Exclusion Criteria:

* Patients with second primary cancer, except:adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumor curatively treated with no evidence of disease for <= 5 years.
* Has known active central nervous system(CNS) metastases
* Has an active infection requiring systemic therapy
* Pregnancy or breast feeding
* Patients with cardiac problem
* Any previous treatment with Sorafenib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | 24 months

SECONDARY OUTCOMES:
Overall Response Rate | 24 months
Time to progression | 24 months
Overall survival | 24 months
Number of subjects with Adverse Events as a measure of safety | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea